CLINICAL TRIAL: NCT00697268
Title: An Investigation to Determine Whether Levels of P11 Protein in Peripheral Blood Cells Correlate With Treatment Response to Citalopram in Patients With Major Depressive Disorder
Brief Title: p11 Protein Levels in Patients With Major Depressive Disorder Treated With Citalopram
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080150; 08-M-0150
Record Dates: First submitted 2008-06-12; First posted 2008-06-13 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-07-28

CONDITIONS: Depression
Keywords: Depression; Depression Treatment; Unipolar Depression; Citalopram; Serotonin; Major Depression; Healthy Volunteer; HV
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major

SUMMARY:
This study will compare levels of p11 protein in people with and without major depressive disorder (MDD) and examine if p11 levels in patients are affected by treatment with citalopram (Celexa).

Healthy normal volunteers and patients with chronic or recurrent major depression between 18 and 65 years of age may be eligible for this study.

Participants undergo the following tests and procedures:

Healthy Volunteers

* Psychiatric interview and medical examination, questions about family history
* Blood draw

Patients with MDD

Phase 1 - Evaluation and Discontinuation of Medications

* Physical examination, electrocardiogram, blood tests
* Gradual antidepressant medication withdrawal, followed by 2- to 6-week drug-free period. If needed, medicines for anxiety and difficulty sleeping may be prescribed.

Phase 2 Citalopram Treatment

* Start daily citalopram treatment
* Evaluations at the start of phase 2 and every week for 8 weeks with following procedures:
* Symptoms ratings interview and questionnaires
* Review of side effects and new medications
* Blood pressure and pulse measurements
* Blood and urine tests

At the end of the study, plans are developed for long-term treatment and transfer of care to the patient s own physician.

...

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a serious, debilitating, life-shortening illness that affects many persons of all ages and backgrounds. While treatments are effective for a significant portion of patients with MDD, progress in developing more effective treatments is lagging. Furthermore, with regards to existing antidepressant medications, there are yet no reliable predictors of the likelihood of remission, response or non-response with an initial trial of an antidepressant medication. Identifying factors that are likely to predict response would have the advantage of personalizing treatment to a particular individual; that is selecting the antidepressant medication that is most likely to give the greatest probability of having a favorable outcome.

The serotonin system has been implicated in the pathophysiology of depression and mechanism of action of existing effective antidepressant treatments. Fourteen different serotonin receptors have been identified to date. One of them, 5-HT1B, plays an important role in regulating serotonin neurotransmission. Recently, p11 (a member of the S100 family of proteins) was found to interact with 5-HT1B receptors (Svenningsson et al 2006; Svenningsson and Greengard 2007). p11 mRNA levels are markedly reduced in the forebrain in helpless H/Rouen mice and the level of p11 mRNA was down-regulated in the anterior cingulate cortex from depressed patients. p11 mRNA is distributed in an anatomical pattern that closely resembled that of 5-HT1B receptor mRNA, including cortex, hippocampus, hypothalamus and raphe nuclei. Chronic administration of the antidepressants imipramine, tranylcypromine, and citalopram significantly increase the level of p11 in cortex. Finally, we have found that chronic treatment with fluoxetine increases p11 in peripheral mononuclear cells in monkeys.

We will now study whether the blood cell levels of p11 differ between healthy individuals and patients suffering from unipolar depression. Moreover, we will study whether the levels of p11 are affected by treatment with the selective serotonin reuptake inhibitor, citalopram. Complementary work will continue at other laboratories to better characterize the role of p11 in the pathophysiology of depression (e.g., animal studies, post-mortem studies).

In addition, we will also acquire a battery of magnetic resonance imaging (MRI) scans in a subset of 45 more homogeneous depressed subjects, and 45 matched healthy controls at baseline and at 8 weeks. There is a growing body of evidence implicating morphometric and physiologic abnormalities, measureable by MRI, in the pathophysiology of major depressive disorder. We will assess both baseline differences between depressed subjects and healthy controls, treatment effects, and search for possible MRI markers predicting treatment response.

This is an open label study which will be performed at the National Institute of Mental Health. In all, 82 adult subjects with major depressive disorder, between the ages of 18 and 65 years, will be recruited from the community. In addition, we will perform p11 measurements in blood cells from 64 healthy control subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

CRITERIA FOR INCLUSION OF DEPRESSED PATIENTS:

* age 18-65 years
* written informed consent completed (consent-incapacitated subjects will not be eligible)
* score 20 or higher on the Montgomery-Asberg Depression Rating Scale (MADRS)
* meets DSM-IV criteria for chronic or recurrent nonpsychotic MDD
* patients who are on non-excluded concomitant medications.
* no more than 3 failed antidepressant treatments within the current major depressive episode
* no alcohol use (last 7 days)

ADDITIONAL CRITERIA FOR INCLUSION OF DEPRESSED PATIENTS FOR MRI IMAGING:

* age 18 55 years
* subjects must have either a family history of mood disorders, or have a history of

multiple major depressive episodes

* age of onset of depressive symptoms less than 45 years
* no history of past alcohol or substance dependence (excluding nicotine) or alcohol or substance abuse (excluding nicotine) within the past year.
* no use of benzodiazepines within 2 weeks of either MRI scan

CRITERIA FOR INCLUSION OF HEALTHY CONTROL SUBJECTS:

* age 18-65 years
* written informed consent completed
* no current or past diagnosis of axis I psychiatric disorder (DSM-IVTR)
* no alcohol use (last 7 days)
* physically healthy

ADDITIONAL CRITERIA FOR INCLUSION OF HEALTHY CONTROL SUBJECTS FOR MRI IMAGING:

* age 18 55 years
* no history of past alcohol or substance dependence (excluding nicotine) or alcohol or substance abuse (excluding nicotine) within the past year.

EXCLUSION CRITERIA:

CRITERIA FOR EXCLUSION OF DEPRESSED PATIENTS:

* history of bipolar disorder (I, II, or NOS) (lifetime)
* history of schizophrenia
* history of schizoaffective disorder or
* psychosis NOS (lifetime)
* history of anorexia nervosa or bulimia nervosa (lifetime)
* current primary obsessive-compulsive disorder (OCD) or current post traumatic stress disorder (PTSD) whose onset preceded the onset of Major Depressive Disorder
* history of clear-cut intolerability to the study medication
* lack of response to an adequate trial of the study medication (citalopram) in the current or past episodes of MDD
* did not respond to 7 or more sessions of ECT in the current episode of MDD
* Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
* has general medical condition which contraindicates the use of the study medication
* is on concomitant medication which contraindicates the use of the study medication
* requires immediate hospitalization for psychiatric disorder
* requires antipsychotic medications or mood stabilizers
* Non-postmenopausal (less than 2 years since last period) females of childbearing potential who are sexually active and who are not using adequate (hormonal, double barrier, surgical) contraception, or who are pregnant or breast feeding
* patients currently taking any of the exclusionary medications detailed in protocol (including antipsychotic medications, anticonvulsant medications, antidepressant medications, mood stabilizers, central nervous system stimulants) in the 2 weeks prior to Study Period II.
* patients taking thyroid medication for hypothyroidism may be included if they have been stable on the medication for greater than 3 months
* patients can participate in a modality of psychotherapy that is not targeting the symptoms of depression (e.g., supportive therapy, marital therapy)
* therapy that is depression specific, such as Cognitive Therapy (CT) or Interpersonal Psychotherapy of Depression (IPT) is not allowed during participation
* subjects must be fluent in English and have the capacity to understand the nature of the study and sign the written informed consent.
* current alcohol dependence or abuse (last 3 months)
* patient has a prolonged QTc (greater than or equal to 450 msec), as shown on ECG
* Current NIMH employee/staff or their immediate family member.

ADDITIONAL CRITERIA FOR EXCLUSION OF DEPRESSED PATIENTS FOR MRI IMAGING:

* subjects meeting general exclusion criteria for MRI scanning (e.g. implanted cardiac pacemaker, intraocular metal) will be excluded from the MRI procedures only.
* subjects with structural lesions visible on MRI will be excluded from further MRI procedures
* subjects with diabetes or hypertension will be excluded

CRITERIA FOR EXCLUSION OF HEALTHY CONTROL SUBJECTS:

* subjects currently taking any of the exclusionary medications detailed in protocol in the 2 weeks prior to evaluation
* current alcohol dependence or abuse (last 3 months)
* history of major depression or bipolar disorder in any first degree relative

ADDITIONAL CRITERIA FOR EXCLUSION OF HEALTHY CONTROL SUBJECTS:

* subjects meeting general exclusion criteria for MRI scanning (e.g. implanted cardiac pacemaker, intraocular metal) will be excluded from the MRI procedures only.
* subjects with structural lesions visible on MRI will be excluded from further MRI procedures
* subjects with diabetes or hypertension will be excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-06-03; Study Completion 2016-07-28

PRIMARY OUTCOMES:
We will study whether blood cell levels of p11 differ between healthy individuals and patients with depression. Moreover, we will study whether the levels of p11 are affected by treatment with the selective serotonin reuptake inhibitor, citalopr... | Baseline, +1 week, +2 weeks, +3 weeks, +4 weeks, +5 weeks, +6 weeks, +7 weeks, +8 weeks

SECONDARY OUTCOMES:
Complementary work will continue at other laboratories to better characterize the role of p11 in the pathophysiology of depression (e.g., animal studies, post-mortem studies). | Baseline, +1 week, +2 weeks, +8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barnes NM, Sharp T. A review of central 5-HT receptors and their function. Neuropharmacology. 1999 Aug;38(8):1083-152. doi: 10.1016/s0028-3908(99)00010-6. PMID 10462127
- [Background] Greenberg PE, Kessler RC, Birnbaum HG, Leong SA, Lowe SW, Berglund PA, Corey-Lisle PK. The economic burden of depression in the United States: how did it change between 1990 and 2000? J Clin Psychiatry. 2003 Dec;64(12):1465-75. doi: 10.4088/jcp.v64n1211. PMID 14728109
- [Background] Katon W, Von Korff M, Lin E, Walker E, Simon GE, Bush T, Robinson P, Russo J. Collaborative management to achieve treatment guidelines. Impact on depression in primary care. JAMA. 1995 Apr 5;273(13):1026-31. PMID 7897786